CLINICAL TRIAL: NCT05287399
Title: An Open-Label, Multicenter, Single-Arm Phase 1 Clinical Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC61 in Subjects With Advanced Solid Tumors
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC61in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASC61-101
Record Dates: First submitted 2022-02-23; First posted 2022-03-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ASC61 200 mg 1 (Experimental): ASC61 200 mg orally once
  Interventions: Drug: ASC61 200 mg 1
- ASC61 200 mg 2 (Experimental): ASC61 200 mg orally twice daily
  Interventions: Drug: ASC61 200 mg 2
- ASC61 300 mg (Experimental): ASC61 300 mg orally twice daily
  Interventions: Drug: ASC61 300 mg
- ASC61 400 mg (Experimental): ASC61 400 mg orally twice daily
  Interventions: Drug: ASC61 400 mg
- ASC61 600 mg (Experimental): ASC61 600 mg orally twice daily
  Interventions: Drug: ASC61 600 mg
- ASC61 800 mg (Experimental): ASC61 800 mg orally twice daily
  Interventions: Drug: ASC61 800 mg

INTERVENTIONS:
Drug: ASC61 200 mg 1 — 200mg of ASC61 orally once daily for cycles of 28 days
  Arms: ASC61 200 mg 1
Drug: ASC61 200 mg 2 — 200 mg of ASC61 orally twice daily for cycles of 28 days
  Arms: ASC61 200 mg 2
Drug: ASC61 300 mg — 300 mg of ASC61 orally twice daily for cycles of 28 days
  Arms: ASC61 300 mg
Drug: ASC61 400 mg — 400 mg of ASC61 orally twice daily for cycles of 28 days
  Arms: ASC61 400 mg
Drug: ASC61 600 mg — 600 mg of ASC61 orally twice daily for cycles of 28 days
  Arms: ASC61 600 mg
Drug: ASC61 800 mg — 800 mg of ASC61 orally twice daily for cycles of 28 days
  Arms: ASC61 800 mg

SUMMARY:
This is a Phase 1, open-label, multicenter, single-arm, dose escalation study, designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of single-agent ASC61(an orally bioavailable small-molecule inhibitor of PD-L1) in subjects with advanced solid tumors for whom no standard therapy is available.

DETAILED DESCRIPTION:
Except for the first starting dose of 200 mg once daily (QD), a traditional "3 + 3 design" will be followed for dose finding with dose escalation and/or de escalation as appropriate. Each subject in each dose cohort will use 2 dose schedules: single dose on Day 1 (D1), and repeated doses on daily basis for 28 days starting from Day 3. One treatment cycle is 28 days. Subjects will be sequentially enrolled in a dose-escalation design to receive ASC61 at initial dose of 200 mg QD. Subsequent doses of 200 mg twice a day (BID), 300 mg BID, 400 mg BID, 600 mg and 800 mg BID are planned.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age at the time of screening
* Histological or cytological diagnosis of advanced/metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available, regardless of cancer stage and previous experienced therapies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least one measurable lesion, as defined by RECIST 1.1

Exclusion Criteria:

* Known symptomatic brain metastases requiring steroids
* Known history of another primary solid tumor
* Subjects discontinued prior therapy with immune checkpoints due to toxicity if previously received therapy with this class of drugs
* Known history of idiopathic pulmonary fibrosis, drug-induced pneumonitis, or evidence of active pneumonia or pneumonitis
* Gastrointestinal disorders that might affect drug absorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience DLTs | From baseline to 28 days of treatment
  The primary endpoint of this study is the proportion of the patients who experience DLTs. The MTD (Maximum Tolerated Dose) will be determined based on the dose escalation cohorts. The evaluation period for DLTs will be 28 days following treatment of PD1-PDL1 inhibitor
Dose(s) of ASC 61 to be examined in Part 2 and the recommended Phase 2 dose(s) | From first dose of ASC61 (Day 1) until 90 days after the last dose
  Maximum serum concentration (Cmax) of ASC61, Area under the serum concentrations of ASC61 versus time curve (AUC) and Half-life (t1/2) of serum concentrations of ASC61)

SECONDARY OUTCOMES:
Percentage of ASC61 subjects with a best response of Complete Response or Partial Response (Objective Response Rate) | Baseline until confirmed disease progression (CR or PR) (up to 1 year)
Percentage of ASC61 subjects with Complete Response, Partial Response, or Stable Disease (Disease Control Rate) | Baseline until confirmed disease progression (CR or PR) (up to 1 year)
Length of time that ASC61 subjects continue to respond to treatment without disease progression (Duration of response) | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (up to 1 year)
Length of time between first dosing and disease progression (Progression-Free survival) | From first dose of ASC61 (Day 1) until death (up to 1 year)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - California Cancer Associates for Research & Excellence (cCARE), Fresno, California
  - California Cancer Associates for Research & Excellence (cCARE), San Marcos, California
  - Nebraska Cancer Specialists, Omaha, Nebraska